CLINICAL TRIAL: NCT04316143
Title: An Open-label, Multicentre Study to Evaluate Pharmacokinetics, Safety and Efficacy of Zamicastat as Adjunctive Therapy in Pulmonary Arterial Hypertension (PAH)
Brief Title: Pharmacokinetics, Safety and Efficacy of BIA 5-1058 in PAH (Zamicastat)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-201; 2018-002448-10 (EudraCT Number)
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; BIA 5-1058; Zamicastat; Bial; Bial - Portela & Ca, S.A.; dopamine ß-hydroxylase (DßH) inhibitor; vascular obstruction; pulmonary arteries; right-heart catheterisation (RHC); idiopathic; rare lung disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 50 mg zamicastat (Experimental): 50 mg zamicastat once daily
  Interventions: Drug: Oral zamicastat
- 100 mg zamicastat once daily (Experimental): 100 mg zamicastat once daily
  Interventions: Drug: Oral zamicastat
- 150 mg zamicastat once daily (Experimental): 150 mg zamicastat once daily
  Interventions: Drug: Oral zamicastat
- 200 mg zamicastat once daily (Experimental): 200 mg zamicastat once daily
  Interventions: Drug: Oral zamicastat

INTERVENTIONS:
Drug: Oral zamicastat — Tablets for oral administration under fed conditions containing 100 mg of zamicastat
  Other Names: BIA 5-1058

SUMMARY:
This Study evaluates the pharmacokinetic (PK) profile of different zamicastat doses in Pulmonary arterial hypertension (PAH) patients to find the most promising therapeutic dosage range for the treatment of PAH disease

DETAILED DESCRIPTION:
This is an open-label, multi-centre study in patients with PAH who are currently on stable treatment with at least one PAH medication. It is planned to evaluate the PK profile (24 hour profile and trough levels) and the safety, tolerability and efficacy of four different zamicastat doses. Each patient will start treatment with the lowest dose (50 mg zamicastat once daily) and the dose will be up-titrated to the individual highest tolerated dose (HTD) i.e. up to 200 mg zamicastat once daily.

A data safety monitoring board (DSMB) will periodically review the safety data and will issue a recommendation if the doses can be used as planned.

This study will consist of:

* A screening period, 5 to 12 days: visit V1
* Up to four dose finding periods, 14 days each:

  * Dose A (50 mg zamicastat once daily): visits A1, A2 and A3
  * Dose B (100 mg zamicastat once daily): visits B2 and B3
  * Dose C (150 mg zamicastat once daily): visits C2 and C3
  * Dose D (200 mg zamicastat once daily): visits D2 and D3
* Maintenance period, 42 days: maintenance period visit (MPV)1, MPV2 and MPV3
* Follow-up (FU) period, 14 to 28 days: visits FU (down-titration) and FU

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 70 years.
2. Able to comprehend and willing to sign an informed consent form.
3. Diagnosis of PAH (pulmonary arterial hypertension WHO Group 1), documented by right heart catheterisation with a mean pulmonary artery pressure (mPAP) ≥ 25 mmHg, a pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg and a pulmonary vascular resistance (PVR) > 3 wood unit (WU):

   1. Idiopathic, in non-vasoreactive patients
   2. Heritable: Bone morphogenetic protein receptor type II (BMPR2) mutation and other mutations, in non-vasoreactive patients
   3. Drugs and toxin induced, in non-vasoreactive patients
   4. Associated with connective tissue disease
   5. Associated with simple congenital defects (atrial septal defect and/or ventricular septal defect) if closed > 12 months before inclusion.
4. World Health Organization (WHO) functional class II or III as judged by the investigator.
5. Stable treatment with at least one of the following approved PAH therapies for at least 90 days prior to V1: Ambrisentan, Bosentan, Macitentan, Riociguat, Selexipag, Sildenafil, Tadalafil, Epoprostenol intravenous, Iloprost inhaled or Treprostinil intravenous or subcutaneous.

Exclusion Criteria:

1. Contraindication to zamicastat, i.e. known hypersensitivity to ingredients of zamicastat formulation.
2. Two or more consecutive measurements of systolic blood pressure (SBP) < 95 mmHg or diastolic blood pressure (DBP) < 50 mmHg.
3. Uncontrolled diabetes mellitus with HbA1c ≥ 8.5% within the last three months or at screening.
4. PAH WHO Group 1 due to portal hypertension, human immunodeficiency virus (HIV) infection and schistosomiasis.
5. Any disease known to cause pulmonary hypertension other than PAH WHO Group 1.
6. Obstructive lung disease: Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) < 60% and FEV1 < 60% of predicted value after bronchodilator administration.
7. Restrictive lung disease: Total Lung Capacity (TLC) < 70% of predicted value.
8. History of moderate to severe hepatic impairment (Child-Pugh B and C).
9. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 (measured at V1).
10. Use of the following prohibited medication or treatments during study participation: calcium channel blockers (CCBs) if used for the treatment of PAH in vasoreactive patients; drugs containing a catechol group that is metabolised by dopamine ß-hydroxylase (DβH) e.g. rimiterole, isoprenaline, dopamine, dopexamine or dobutamide or α- and/or β-blockers.
11. Current or previous (within the past year) alcohol or substance abuse excluding caffeine or nicotine.
12. Presence of any other significant or progressive/unstable medical condition that, in the opinion of the investigator, would compromise evaluation of the study treatment or may jeopardise the patient's safety, compliance or adherence to protocol requirements.
13. For women: Pregnancy or breast-feeding. Women of childbearing potential unable or unwilling to undergo pregnancy tests and practice acceptable contraceptive measures from the time of informed consent until 30 days after last investigational medicinal product (IMP) intake. Acceptable methods for women are surgical intervention (e.g. bilateral tubal occlusion), non-hormonal implantable intrauterine device, double-barrier methods, true sexual abstinence (i.e. when this is in line with the preferred and usual lifestyle of the patient) and vasectomised partner (provided that the partner is the sole sexual partner of the patient and the partner has received medical assessment of the surgical success). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), hormonal contraceptives and withdrawal are not acceptable methods of contraception.

    For men: Male patients who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved acceptable contraceptive measure from the time of informed consent until 90 days after the last IMP intake. The following methods are acceptable methods of contraception: partner's use of combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); partner's use of progestogen-only hormonal contraception (oral, injectable/implantable, intrauterine hormone-releasing system); partner's use of implantable intrauterine device; surgical sterilisation (for example, vasectomy or bilateral tubal occlusion).
14. Previous participation in any other drug investigational study within the past 30 days (or five half-lives of IMP whichever is longer) prior to V1.
15. Vulnerable patients according to Section 1.61 of the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guideline for Good Clinical Practice E6.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Ordensklinikum Linz Elisabethinen, Interne 2 - Kardiologie, Angiologie & Interne Intensivmedizin Fadingerstraße 1, Linz, Austria
- Universitätsklinikum Carl Gustav Carus Dresden, Medizinische Klinik und Poliklinik I, Pneumologie Fetscherstraße 74, Dresden, Germany
- Italy (3):
  - Ospedale Generale Regionale Miulli-Cardiologia e UTIC Strada Prov. 127 Acquaviva - Santeramo Km. 4,100, Acquaviva delle Fonti
  - ASST di Monza-Ospedale San Gerardo -Dipartimento di Pneumologia via Pergolesi 33, Monza
  - AOU di Roma-Policlinico Umberto I-Unità Dipartimentale Malattie del Circolo Polmonare Viale del Policlinico 155, Roma
- Centro Hospitalar Lisboa Norte, E.P.E. - Hospital Pulido Valente Consulta Externa de Hipertensão Pulmonar Alameda das Linhas de Torres, 117, Lisbon, Portugal
- Spain (4):
  - Hospital Clinic de Barcelona Calle Villarroel, 170, Barcelona
  - Hospital Universitario "12 de Octubre" Avda. de Córdoba, s/n, Madrid
  - Complejo Asistencial Universitario de Salamanca Pº. San Vicente, 58, Salamanca
  - Hospital Universitario Marques de Valdecilla Avenida Valdecilla, 25, Santander
- State Institution ""National Scientific Centre "M.D. Strazhesko Institute of Cardiology" of NAMS of Ukraine", Department of symptomatic arterial hypertensions Narodnogo opolcheniya 5, Kyiv, Ukraine
- United Kingdom (2):
  - Golden Jubilee National Hospital Golden Jubilee National Hospital Agamemnon St, Scottish Pulmonary Vascular Unit Golden Jubilee National Hospital, Clydebank
  - Royal Free Hospital Pond Street, London

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 33 patients enrolled in this study, 29 patients started treatment with zamicastat (4 Screening Failures), 28 patients completed the dose finding period and entered the maintenance period (1 premature termination). Patients who had been enrolled and, for whatever reason, discontinued the study after first IMP intake at visit A1 were classified as withdrawals. Patients might withdraw from the study at any time, either on their own request or at the discretion of the investigator.
Groups:
- 50 mg Zamicastat: 50 mg zamicastat once daily (half a tablet of 100 mg)
  Zamicastat: Tablets for oral administration under fed conditions containing 100 mg of zamicastat (BIA 5-1058)
- 100 mg Zamicastat Once Daily: 100 mg zamicastat once daily (one tablet of 100 mg)
  Zamicastat: Tablets for oral administration under fed conditions containing 100 mg of zamicastat (BIA 5-1058)
- 150 mg Zamicastat Once Daily: 150 mg zamicastat once daily (one and a half tablet of 100 mg)
  Zamicastat: Tablets for oral administration under fed conditions containing 100 mg of zamicastat (BIA 5-1058)
- 200 mg Zamicastat Once Daily: 200 mg zamicastat once daily (two tablets of 100 mg)
  Zamicastat: Tablets for oral administration under fed conditions containing 100 mg of zamicastat (BIA 5-1058)
Period: 50 mg Toleration Period - Dose A
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Started | 29 (If dose has been tolerated during 14-day treatment, up-titrate to Dose B, if not withdraw patient) | 0 | 0 | 0
Completed | 27 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Period: 100 mg Toleration Period - Dose B
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Started | 0 | 27 (If dose has been tolerated during 14-day treatment, up-titrate to Dose C, if not withdraw patient) | 0 | 0
Completed | 0 | 21 | 0 | 0
Not Completed | 0 | 6 | 0 | 0
Period: 150 mg Toleration Period - Dose C
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Started | 0 | 0 | 21 (If dose has been tolerated during 14-day treatment, up-titrate to Dose D, if not withdraw patient) | 0
Completed | 0 | 0 | 19 | 0
Not Completed | 0 | 0 | 2 | 0
Period: 200 mg Toleration Period - Dose D
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Started | 0 | 0 | 0 | 19
Completed | 0 | 0 | 0 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily | Total
Number analyzed (Participants) | 1 | 6 | 2 | 19 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 6 | 2 | 16 | 25
  >=65 years | 0 | 0 | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 14 | 21
  Male | 0 | 1 | 1 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 6 | 2 | 19 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height (cm) [Count of Participants; unit: Participants] — Category title defined according Median presented in Table 15.1.6.2.2 Baseline Characteristics - Full Analysis Set
  Participants
    <=1.65cm | 0 | 1 | 0 | 12 | 13
    >1.65 | 1 | 5 | 2 | 7 | 15
Weight (kg) [Count of Participants; unit: Participants] — Category title defined according Median presented in Table 15.1.6.2.2 Baseline Characteristics - Full Analysis Set
  Participants
    <71,5kg | 0 | 3 | 1 | 16 | 20
    >71,5kg | 1 | 3 | 1 | 3 | 8
BMI (kg/m2) [Count of Participants; unit: Participants] — Category title defined according Median presented in Table 15.1.6.2.2 Baseline Characteristics - Full Analysis Set
  Participants
    <=25,4kg/m2 | 0 | 4 | 2 | 9 | 15
    >=25,5kg/m2 | 1 | 2 | 0 | 10 | 13
Childbearing Potential [Count of Participants; unit: Participants]
  Yes | 0 | 4 | 1 | 6 | 11
  No | 1 | 2 | 0 | 8 | 11
  Not Applicable | 0 | 0 | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0-24h (AUC0-24h) (ng.h/mL) - 50 mg
Description: This PK parameters (24-hour profile) for zamicastat and its metabolites will be derived after a single dose of 50 mg zamicastat
Time Frame: Day 1 (0 hours and then 1, 2, 4, 8, 16 and 24 hours after investigational medicinal product (IMP) intake)
Population: Following multiple administrations of the HTD of zamicastat to pulmonary arterial hypertension (PAH) patients at maintenance period visit (MPV)3, pharmacokinetic (PK) concentrations and parameter summaries for only the 50 mg, 100 mg and 200 mg dose levels are presented and discussed, as the only subject receiving the 150 mg HTD level had a major protocol deviation documented, impacting the reliability of their PK data.
Measure: Geometric Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Number analyzed (Participants) | 1 | 4 | 0 | 17
ng.h/mL
  Zamicastat | 155 | 761 (44.6) |  | 1570 (59.7)
  BIA 5-453_1: number analyzed (Participants) | 0 | 1 | 0 | 14
  BIA 5-453_1 |  | 172 |  | 305 (38.5)
  BIA 5-453_2: number analyzed (Participants) | 0 | 1 | 0 | 14
  BIA 5-453_2 |  | 181 |  | 305 (38.5)
  BIA 5-961: number analyzed (Participants) | 0 | 2 | 0 | 15
  BIA 5-961 |  | 150,187 (0) |  | 277 (94.3)

2. Primary Outcome: Area Under the Curve 0-24h (AUC0-24h) (ng.h/mL/mg) - HTD
Description: This PK parameter (24-hour profile) for zamicastat and its metabolites will be derived at steady-state at the individual highest tolerated dose (HTD)
Time Frame: 1, 2, 4, 8, 16 and 24 hours after IMP intake
Population: Following multiple administrations of the HTD of zamicastat to PAH patients at MPV3, PK concentrations and parameter summaries for only the 50 mg, 100 mg and 200 mg dose levels are presented and discussed, as the only subject receiving the 150 mg HTD level had a major protocol deviation documented, impacting the reliability of their PK data.
Measure: Geometric Mean (Standard Deviation); unit: ng.h/mL/mg
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Number analyzed (Participants) | 1 | 4 | 0 | 17
ng.h/mL/mg
  Zamicastat | 3.09 | 7.61 (44.6) |  | 7.87 (59.7)
  BIA 5-453_1: number analyzed (Participants) | 0 | 1 | 0 | 14
  BIA 5-453_1 |  | 1.72 (0) |  | 1.53 (38.5)
  BIA 5-453_2: number analyzed (Participants) | 0 | 1 | 0 | 14
  BIA 5-453_2 |  | 1.81 |  | 1.53 (38.5)
  BIA 5-961_1: number analyzed (Participants) | 0 | 1 | 0 | 15
  BIA 5-961_1 |  | 1.50 |  | 1.39 (94.3)
  BIA 5-961_2: number analyzed (Participants) | 0 | 1 | 0 | 15
  BIA 5-961_2 |  | 1.87 |  | 1.39 (94.3)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) (ng/mL) - 50 mg
Description: as for outcome 1
Time Frame: Day 1 (0 hours and then 1, 2, 4, 8, 16 and 24 hours after IMP intake)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Number analyzed (Participants) | 1 | 4 | 0 | 17
ng/mL
  Zamicastat | 13.3 | 62.6 (60.5) |  | 134 (94.0)
  5-453: number analyzed (Participants) | 0 | 4 | 0 | 15
  5-453 |  | 8.39 (33.1) |  | 18.8 (48.1)
  BIA 5-961_1: number analyzed (Participants) | 1 | 1 | 0 | 17
  BIA 5-961_1 | 5.39 | 11.0 |  | 17.6 (78.2)
  BIA 5-961_2: number analyzed (Participants) | 1 | 1 | 0 | 17
  BIA 5-961_2 | 5.39 | 23.9 |  | 17.6 (78.2)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) (ng/mL/mg) - HTD
Description: as for outcome 2
Time Frame: 1, 2, 4, 8, 16 and 24 hours after IMP intake
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Number analyzed (Participants) | 1 | 4 | 0 | 17
ng/mL/mg
  Zamicastat | 0.27 | 0.626 (60.5) |  | 0.672 (94.0)
  BIA 5-453: number analyzed (Participants) | 0 | 4 | 0 | 15
  BIA 5-453 |  | 0.0839 (33.1) |  | 0.0939 (48.1)
  BIA 5-961_1: number analyzed (Participants) | 1 | 1 | 0 | 17
  BIA 5-961_1 | 0.108 | 0.110 |  | 0.0882 (78.2)
  BIA 5-961_2: number analyzed (Participants) | 1 | 1 | 0 | 17
  BIA 5-961_2 | 0.108 | 0.239 |  | 0.0882 (78.2)

5. Primary Outcome: Time Until Cmax (Tmax) (h) - 50 mg
Description: as for outcome 1
Time Frame: Day 1 (0 hours and then 1, 2, 4, 8, 16 and 24 hours after IMP intake)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Number analyzed (Participants) | 1 | 4 | 0 | 17
h
  Zamicastat | 2.00 | 3.00 (1.00) |  | 4.00 (1.00)
  BIA 5-453: number analyzed (Participants) | 0 | 4 | 0 | 15
  BIA 5-453 |  | 3.00 (2.00) |  | 4.05 (2.00)
  BIA 5-961: number analyzed (Participants) | 1 | 1 | 0 | 17
  BIA 5-961 | 4.03 | 2.00 |  | 8.00 (4.00)

6. Primary Outcome: Time Until Cmax (Tmax) (h) - HTD
Description: as for outcome 2
Time Frame: 1, 2, 4, 8, 16 and 24 hours after IMP intake
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Number analyzed (Participants) | 1 | 4 | 0 | 17
h
  Zamicastat | 2.00 | 3.00 (4.08) |  | 4.00 (24.00)
  BIA 5-453: number analyzed (Participants) | 0 | 4 | 0 | 15
  BIA 5-453 |  | 3.00 (8.08) |  | 4.05 (24.0)
  BIA 5-961: number analyzed (Participants) | 1 | 1 | 0 | 17
  BIA 5-961 | 4.03 | 8.08 |  | 8.00 (24.0)

7. Primary Outcome: Minimum Plasma Concentration at the End of the Dosing Interval (Cmin,SS) (ng/mL/mg) - HTD
Description: This PK parameter (24-hour profile) for zamicastat and its metabolites will be derived at steady-state at the individual highest tolerated dose (HTD). Following multiple administrations of the HTD of zamicastat to PAH patients at MPV3, PK concentrations and parameter summaries for only the 50 mg, 100 mg and 200 mg dose levels are presented and discussed, as the only subject receiving the 150 mg HTD level had a major protocol deviation documented, impacting the reliability of their PK data.
Time Frame: 1, 2, 4, 8, 16 and 24 hours after IMP intake
Population: Non-numerical values reported in the plasma concentration data (i.e. values that are below the limit of quantification), will be treated as missing for the determination of summary statistics. This also applies to any concentrations that are defined as PK parameters (e.g. Cmin). Where less than 3 patients receive the same dose at MPV3 or there are less than 3 quantifiable concentrations at a time point or parameter, summary statistics will not be produced for this dose/visits or time point.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
Number analyzed (Participants) | 1 | 4 | 0 | 17
ng/mL/mg
  Zamicastat: number analyzed (Participants) | 0 | 4 | 0 | 17
  Zamicastat |  | 0.186 (36.7) |  | 0.198 (74.1)
  BIA 5-453_1: number analyzed (Participants) | 0 | 1 | 0 | 14
  BIA 5-453_1 |  | 0.0564 |  | 0.0479 (48.5)
  BIA 5-453_2: number analyzed (Participants) | 0 | 1 | 0 | 14
  BIA 5-453_2 |  | 0.0603 |  | 0.0479 (48.5)
  BIA 5-961: number analyzed (Participants) | 0 | 1 | 0 | 14
  BIA 5-961 |  | 0.0896 |  | 0.0503 (58.6)

ADVERSE EVENTS:
Time Frame: 94,5 days
Description: In the overall population, 23 (79.3%) patients experienced 94 TEAEs during the study. The overall frequency of TEAEs was comparable between patients taking 100mg (15 patients, 53.6%), 150mg (15 patients, 55.6%) and 200mg (11 patients, 52.4%) doses at onset of TEAEs, whereas the lowest frequency (10 patients, 34.5%) was observed for patients receiving 50mg. Most TEAEs (68 out of 94) were assessed as mild in intensity, 26 TEAEs were assessed as moderate in intensity. No severe TEAEs were reported.
Arm/Group | 50 mg Zamicastat | 100 mg Zamicastat Once Daily | 150 mg Zamicastat Once Daily | 200 mg Zamicastat Once Daily
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28 | 0/27 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/28 | 0/27 | 0/21
Other Adverse Events (participants affected / at risk) | 10/29 | 15/28 | 15/27 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Zamicastat (N=29) | 100 mg Zamicastat Once Daily (N=28) | 150 mg Zamicastat Once Daily (N=27) | 200 mg Zamicastat Once Daily (N=21)
Device breakage (Product Issues) | 0 | 1 | 0 | 0 — Possible Hickman line fracture
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Clinical worsening of PAH
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Zamicastat (N=29) | 100 mg Zamicastat Once Daily (N=28) | 150 mg Zamicastat Once Daily (N=27) | 200 mg Zamicastat Once Daily (N=21)
Ventricular extrasystoles (Cardiac disorders) | 0 | 2 | 0 | 0 — VENTRICULAR EXTRASYSTOLES
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 2 | 1 — RESPIRATORY ARRHYTHMIA
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 — NAUSEA
Fatigue (General disorders) | 1 | 1 | 2 | 1 — FATIGUE
Feeling abnormal (General disorders) | 0 | 1 | 1 | 0 — FOGGY-HEADEDNESS
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — JAW PAIN
Syncope (Nervous system disorders) | 0 | 1 | 1 | 1 — SYNCOPE
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — CUTANEOUS HYPERSENSITIVITY
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — EXANTHEMA
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0 — HYPOTENSION
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 — ORTHOSTATIC HYPOTENSION
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 0 — COLD
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 — UPPER RESPIRATORY TRACT INFECTION
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 — TONSILLITIS
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 — HEADACHE
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 — HERPES SIMPLEX
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 — GASTROINTESTINAL INFECTION
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 — VIROSIS
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 — DIZZINESS WORSENING LIGHTHEADEDNESS
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 — ABDOMINAL PAIN
Pyrexia (General disorders) | 1 | 0 | 0 | 0 — FEVER
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0 — CIRCULATORY DYSREGULATION
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — TEMPOROMANDIBULAR PAIN
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 — DYSMENORRHEA
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 — PRE-SYNCOPE
Sleep deficit (Nervous system disorders) | 0 | 1 | 0 | 0 — LACK OF SLEEP
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 — DIARRHOEA
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — WORSENING OF DIVERTICULOSIS
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 — ALT INCREASE
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 — GAMMA-GLUTAMYLTRANSFERASE INCREASE
International normalised ratio abnormal (Investigations) | 0 | 1 | 0 | 0 — ALTERED INR
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 — PALLOR
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 1 — INSOMNIA
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 — WORSENING OF THE DEPRESSIVE SYNDROME
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — THROMBOCYTOPENIA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — HYPERKALAEMIA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — HYPERTRIGLYCERIDEMIA
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — CLINICAL WORSENING OF PAH
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — PAH WORSENING
Device breakage (Product Issues) | 0 | 1 | 0 | 0 — POSSIBLE HICKMAN LINE FRACTURE
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — WORSENING GASTROESOPHAGEAL REFLUX DISEASE
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — VOMITING
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 — AST INCREASE
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 — INCREASING OF GLUCOSE
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0 — FERROPENIA
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — PAPULAR RASH
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0 — LOW ATRIAL RHYTHM
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 — BACK PAIN
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — HYPEREOSINOPHILIA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — LYMPHOCYTIC LEUKOPENIA
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 — INTERMITTENT MICROSCOPIC HAEMATURIA
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 — RENAL DYSFUNCTION
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — EPIGASTRIC PAIN
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — IRRITABLE COLON WORSENING
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — TOOTH PAIN
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 — CRP VALUE INCREASE
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 — FACE HEMATOMA
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 — ANXIETY
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — SKIN LESIONS
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — LOWER LIMB MUSCULAR PAIN WHILE WALKING
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — WORSENING OF DIABETES MELLITUS
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — WORSENING SHORTNESS OF BREATH
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 1 — GALLBLADDER POLYPS
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — SWEATING

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT04316143/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04316143/SAP_001.pdf
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT04316143/ICF_002.pdf